CLINICAL TRIAL: NCT04145622
Title: Phase I/II, Two-Part, Multicenter First-in-Human Study of Ifinatamab Deruxtecan (DS-7300a, I-DXd) in Subjects With Advanced Solid Malignant Tumors (IDeate-PanTumor01)
Brief Title: Study of Ifinatamab Deruxtecan (DS-7300a, I-DXd) in Participants With Advanced Solid Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS7300-A-J101; 194992 (Other: JapicCTI)
Record Dates: First submitted 2019-10-17; First posted 2019-10-30 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Malignant Solid Tumor
Keywords: Advanced Solid Tumor; Malignant Tumor; Ifinatamab deruxtecan (I-DXd)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): Participants with advanced solid tumors who received I-DXd IV Q3W monotherapy during dose escalation phase. Enrollment to this phase is currently closed.
  Interventions: Drug: Ifinatamab deruxtecan (I-DXd)
- Dose expansion (Experimental): Currently enrolling participants with advanced solid tumors who will receive I-DXd IV Q3W monotherapy at the recommended dose for expansion.
  Interventions: Drug: Ifinatamab deruxtecan (I-DXd)

INTERVENTIONS:
Drug: Ifinatamab deruxtecan (I-DXd) — A total anti-B7H3 antibody and MAAA-1181a

SUMMARY:
This is a single group study of participants with advanced solid tumors who have not been cured by other treatments. It is the first time the drug will be used in humans, and will be in two parts.

The primary purpose of the parts are:

* Dose Escalation Part: To evaluate the safety and tolerability and to determine the maximum tolerated dose and the recommended dose for expansion of ifinatamab deruxtecan (I-DXd).
* Dose Expansion Part: To investigate the safety, tolerability and antitumor activity of I-DXd when administered as a single agent.

This study is expected to last approximately 5 years from the time the first participant is enrolled to the time the last participant is off the study.

The number of treatment cycles is not fixed in this study. Participants who continue to benefit from the study treatment may continue, unless:

* they withdraw
* their disease gets worse
* they experience unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Has at least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 on computed tomography (CT) or magnetic resonance imaging (MRI) as assessed by Investigator. Measurable lesions should not be from a previously irradiated site. If the lesion at a previously irradiated site is the only selectable target lesion, a radiological assessment showing significant progression of the irradiated lesion should be provided by the Investigator
* Has adequate cardiac, hematopoietic, renal and hepatic functions
* Has an adequate treatment washout period prior to start of study treatment
* Has a pathologically documented advanced/unresectable or metastatic head and neck squamous cell carcinoma, esophageal squamous cell carcinoma, squamous and adenocarcinoma non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), bladder cancer, sarcoma, endometrial cancer, melanoma, adenocarcinoma CRPC (primary neuroendocrine or histologically confirmed neuroendocrine differentiated prostate cancer is not allowed), breast cancer that is refractory to or intolerable with standard treatment, or for which no standard treatment is available.

For Expansion Cohort 4 2L ESCC participants only:

* Has disease progression a post platinum-based and an immune checkpoint inhibitor (ICI) treatment per global or local guidelines, with a maximum of one prior line of systemic therapy for unresectable advanced or metastatic ESCC.

Exclusion Criteria:

* Has prior treatment with B7-H3 targeted agent, including I-DXd.
* Has had prior discontinuation of an antibody drug conjugate (ADC) that consists of an exatecan derivative (e.g., trastuzumab deruxtecan) due to treatment-related toxicities.
* Has multiple primary malignancies within 3 years, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, superficial GI tract tumors and non-muscle invasive bladder cancer curatively resected by endoscopic surgery.
* Uncontrolled significant cardiovascular disease
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder, or any autoimmune, connective tissue or inflammatory disorders with potential pulmonary involvement, prior pneumonectomy, or requirement for supplemental oxygen
* Has an uncontrolled infection requiring systemic therapy.
* Has substance abuse or any other medical conditions that would increase the safety risk to the subject or interfere with participation of the subject or evaluation of the clinical study in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-11-03 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence of dose-limiting toxicities (DLTs) | Day 1 to Day 21 in Cycle 1 in the dose escalation part
Evaluate the incidence of adverse events (AEs) | Cycle 1 Day 1 through disease progression within 8 cycles (each cycle is 21 days)
Investigate the antitumor activity of ifinatamab deruxtecan (I-DXd) | Cycle 1 Day 1 through disease progression within 8 cycles (each cycle is 21 days)

SECONDARY OUTCOMES:
Characterize the PK parameter AUClast | Cycle 1 Day 1 through disease progression within 8 cycles (each cycle is 21 days)
Characterize the PK parameter AUCtau | Cycle 1 Day 1 through disease progression within 8 cycles (each cycle is 21 days)
Characterize the PK parameter Cmax | Cycle 1 Day 1 through disease progression within 8 cycles (each cycle is 21 days)
Characterize the PK parameter Tmax | Cycle 1 Day 1 through disease progression within 8 cycles (each cycle is 21 days)
Characterize the PK parameter Ctrough | Cycle 1 Day 1 through disease progression within 8 cycles (each cycle is 21 days)
Assess the incidence of anti-drug antibodies (ADAs) | Cycle 1 Day 1 through disease progression within 8 cycles (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (25):
- United States (15):
  - Cedars-Sinai Medical Center- Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Orlando, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Sidney Kimmel Cancer Center - Thomas Jefferson, Philadelphia, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - MDACC (MD Anderson Cancer Center), Houston, Texas
- Japan (10):
  - Aichi Cancer Center Hospital, Aichi
  - National Cancer Center Hospital East, Chiba
  - Hokkaido University Hospital, Hokkaido
  - Osaka University Hospital, Osaka
  - Kindai University Hospital, Ōsaka-sayama
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center Hospital and Research Institute, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - Cancer Institute Hospital of JFCR, Tokyo
  - Showa University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/